CLINICAL TRIAL: NCT01336478
Title: Safety and Toxicity of Escalating Doses of Adoptively Infused ex Vivo Selected CD56+CD3- NK Cells on Day 7 Following Allogeneic Stem Cell Transplantation in Patients With Hematological Malignancies.
Brief Title: CD56+CD3- NK Cells Following Allogeneic Stem Cell Transplantation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JROHH0203
Record Dates: First submitted 2011-03-22; First posted 2011-04-18 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2012-03

CONDITIONS: Haematological Malignancies; Allogeneic Stem Cell Transplant; CD56+CD3- NK Cells
Keywords: NK; natural killer; immunotherapy; leukemia; hematological malignancies; stem cell transplantation; adoptive therapy
MeSH Terms: conditions — Leukemia; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Infusion of donor derived ex-vivo selected NK cells to patients after transplant — Infusion of donor derived ex-vivo selected NK cells to patients after transplant
Procedure: Haematology / Blood chemistry sampling — Haematology / Blood chemistry sampling, collection of blood for ancillary lab research

SUMMARY:
The investigators propose a nonrandomized, Phase I study to assess the safety of infusion of NK cells that will be selected from sibling donors and infused to patients with hematological malignancies early following allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HSCT) is a very effective treatment for a number of hematological malignancies but relapse remains a major problem, especially in patients with high risk disease. Natural killer (NK) cells are immune cells that recognize and kill virally infected cells and tumor cells. NK cells are identified by the expression of the CD56 surface antigen and the lack of CD3. Their ability to kill tumor cells makes them promising to evaluate as effector cells for immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing an allogeneic HSCT from a sibling donor, as treatment for a hematological malignancy. The conditioning regimen, and in particular whether ablative or non ablative, will not be considered in the criteria for recruitment
2. Patient and donor Age >18 years
3. Patients and donors must have signed an informed consent form
4. The donor must be willing and capable of donating lymphocytes for NK selection using apheresis techniques
5. Donor must be fit to undergo leukapheresis

Exclusion Criteria:

1. Life expectancy < 3 months
2. ECOG performance status 3 or 4
3. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, life threatening cardiac arrhythmia
4. Patients will not be eligible if they receive in vivo T depletion with ATG, ALG or campath-1H
5. HIV-positive patients
6. Psychiatric illness/social situations that would limit compliance with study requirements and ability to comprehend the investigational nature of the study and provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Safety and toxicity donor CD56+CD3- NK cells | Day 28 post NK cell infusion
  To evaluate the safety and toxicity of escalating doses of ex vivo selected donor CD56+CD3- NK cells, adoptively infused on day 7 following sibling allogeneic stem cell transplantation in patients with hematological malignancies. We will specifically look for the proportion of patients who develop infusion related toxicity. Toxicity will be defined as per the Common Terminology Criteria for Adverse Events v3.0 (CTCAE).

SECONDARY OUTCOMES:
Donor neutrophil and platelet engraftment | Day 28 post stem cell infusion
  Donor neutrophil engraftment (Neut > 0.5 x10^9/L) and platelet engraftment (Plt > 20 x10^9/L)
Rates of acute GVHD (grade 2-4) | Day 100 post stem cell infusion
  Risk of acute GVHD
Relapse rate | 1 year post stem cell infusion
  Relapse

CONTACTS AND LOCATIONS:
Overall Officials: Katy Rezvani, MD, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Hammersmith Hospital, London, United Kingdom